CLINICAL TRIAL: NCT02086422
Title: Iatrogenic Chronotropic Incompetence and Exercise Tolerance in Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CD13/10799
Record Dates: First submitted 2013-11-26; First posted 2014-03-13 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Heart Failure
MeSH Terms: interventions — Ivabradine; Exercise

ARMS (2):
- ivabradine (Active Comparator): Exercise with ivabradine
  Interventions: Drug: ivabradine; Other: Exercise
- Placebo (Placebo Comparator): Exercise with placebo
  Interventions: Drug: Placebo; Other: Exercise

INTERVENTIONS:
Drug: ivabradine
  Arms: ivabradine
Drug: Placebo
  Arms: Placebo
Other: Exercise

SUMMARY:
Patients with CHF benefit from heart rate lowering, and the investigators have previously demonstrated that this does not adversely affect exercise tolerance. In a pacemaker population we also have shown that preventing heart rate lowering is detrimental in terms of symptoms and prognosis.

The aim of the study is to therefore to establish whether heart rate limitation in patients with heart failure has a negative impact on exercise capacity. If the investigators establish that this is not the case, physicians will be able to confidently prescribe heart rate lowering agents, and programme pacemakers to allow bradycardia without the concern that there will be detrimental effects of symptom.

ELIGIBILITY:
Inclusion Criteria:

* Able to walk on a treadmill Able to provide consent Heart failure (or not) depending upon the arm. Patients with atrial fibrillation to have had an AV node ablation (or very slow response to AF)

Exclusion Criteria:

* Cognitive impairment, known reaction to ivabradine, musculoskeletal issues limiting walking on a treadmill.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2013-07; Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Examining the effects of iatrogenic CI on exercise capacity | 24 months
  Each subject will undergo a full echocardiographic examination.We will assess LV systolic and diastolic function variables, mitral regurgitation, and pulmonary artery pressure.

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom